CLINICAL TRIAL: NCT00988299
Title: Energy Expenditure Responses to Acute Exercise in Older Women
Brief Title: Energy Expenditure Responses to Acute Exercise in Older Women (Calorie Expenditure and Exercise)
Acronym: CEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 09-0864; K99AG031297 (NIH)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Aging
Keywords: older; NEAT; exercise; RMR; energy expenditure
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: exercise — exercise sessions at 45% and 60% of maximum effort

SUMMARY:
In older, normal-weight women (60-75 yrs, BMI=18-28 kg/m2), an acute bout of higher-intensity (60% of maximum effort) aerobic exercise, in comparison to an isocaloric bout of lower-intensity (45% of maximum effort) exercise (caloric expenditure of 3.5 kcal/kg body weight for both), will result in differential:

1. decline in non-exercise activity calorie expenditure in the subsequent 48 hours after exercise;
2. increase in resting metabolic rate 48 hours after exercise;
3. increase in serum free triiodo-L-thyronine (free T3) concentrations immediately following exercise;
4. decline from pre-exercise in plasma leptin and serum free T3 concentrations 48 hours after exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Women
2. Age 60-75 years
3. normal weight
4. Weight-stable (± 5%) within the previous 3 months
5. Non-smoking for last year
6. Able to provide own transportation to study visits
7. Not currently involved in any other research study
8. Willing and able to participate in all aspects of the trial including research testing
9. Willing to give informed consent to participate

Exclusion Criteria:

1. Self-reported significant cardiovascular disease
2. Other self-reported medical conditions such as diabetes, chronic or recurrent respiratory conditions, active cancer, musculoskeletal disease
3. Medications known to affect exercise performance or metabolism
4. Excess caffeine use (> 500mg/day)
5. Any self-reported contraindications to exercise
6. Clinical depression
7. Abnormal cognitive function -

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
non-exercise activity calorie expenditure | 2 days after exercise sessions

SECONDARY OUTCOMES:
resting metabolic rate | 2 days after exercise sessions

CONTACTS AND LOCATIONS:
Overall Officials: Xuewen Wang, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States